CLINICAL TRIAL: NCT04705649
Title: Tailored Adjuvant Therapy in POLE-mutated and p53-wildtype Early Stage Endometrial Cancer
Acronym: TAPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Jessica McAlpine, Gynaecologic Oncologist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAPER
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment de-escalation — De-escalation from standard treatment based on molecular profile

SUMMARY:
Endometrial cancer(EC) is the 4th most common cancer in women globally. Clinicians struggle to determine 'the best' treatment for endometrial cancers as they are very hard to tell apart under the microscope. Our BC team developed and validated a low-cost practical tool that can reliably distinguish ECs by molecular features. Molecular classification can inform women about the likelihood of their disease coming back as well as which treatments might work best for them or are not needed. Investigators are studying how this classifier can identify women at very low risk of disease recurrence in order to spare them toxic therapies.

DETAILED DESCRIPTION:
Purpose:

This proposal will for the first time test the clinical utility of ProMisE in a pan-Canadian setting. Through molecular classification, Investigators are closer to providing consistent treatment to women with EC reducing disparities in care as might be observed according to geography/access to care, and/or racial differences. As the primary focus for this trial investigators will focus on identifying women investigators believe may be overtreated, working to avoid giving toxic therapies with consequential side effects of treatment as many women with EC may be cured by surgery alone. However, by performing molecular classification for all new ECs enrolled investigators will also be able to identify women who are at increased risk of recurrence or death from their disease based on molecular features and direct them to molecular-subtype-specific clinical trials. This will, investigators believe, reduce undertreatment (not identifying and treating women at high risk for recurrence) and will help select the best treatment according to an individuals tumor biology. In summary, the research proposed will assess the feasibility and impact of ProMisE-directed care within a rigorous clinical setting - fulfilling the last step in bringing molecular classification-driven care to women across the country with EC and ultimately improving outcomes for women with this disease.

Hypothesis:

There is a subgroup of early stage endometrial carcinomas that are at very low risk of pelvic recurrence and can be identified through molecular classification providing an opportunity to withhold or deescalate adjuvant therapy.

Objectives:

Primary Objective:

Determine if women with POLE-mutated or p53 wild type/NSMP early stage endometrial cancer who undergo surgery (hysterectomy, BSO, +/-LND)have a low risk (<5%) risk of pelvic (including vaginal) recurrence at 3 years with no or de-escalated adjuvant treatment.

Secondary Objectives:

1. Determine recurrence-free survival.
2. Determine overall survival.
3. Determine sites of recurrence (vaginal, pelvic, distant).
4. Determine health economic impact of molecular classification-tailored adjuvant therapy on the cost of treating endometrial cancer
5. Determine the impact of molecular classification on patient Decisional Conflict Scale (DCS)
6. Determine if variability in adjuvant treatment given to women with endometrial cancer is decreased by molecular classification-tailored adjuvant therapy as compared to current/historic standard of care.

Exploratory Objectives:

1. Are there additional molecular parameters that further stratify risk of recurrence within POLE or p53wt ECs.

Other mutations are also on the Contextual Genomics FindIt™ panel and will be recorded for testing of prognostic or predictive value but will not be used to stratify care nor direct therapy in real time. Similarly L1CAM IHC on whole sections of representative tumor will be performed and tested for associations with outcomes. Additional analysis might include further IHC, proteomic, epigenetic assessment, and immune markers.Investigators will have the opportunity to weigh multiple molecular and clinicopathological parameters captured in data collection post hoc to see if any of these improve prognostic ability when applied with ProMisE.

Research design:

This is A single arm prospective cohort study is the most efficient trial design to address the primary hypothesis. Study investigators have experience with similar successful trials in other disease sites (breast-DUCHESS, LUMINA). Some components of this molecular based tool are now widely reported on standard of care pathology reports (MMRd, p53) making the possibility of creating a cohort blinded to these molecular results and thus randomization of this cohort impractical. With implications of these molecular features impacting HCP referrals, pathology categorization, and treatment opportunities (e.g., immune blockade) it is not appropriate to withhold these molecular results from patients. Randomization and creation of true blinded cohorts are therefore no longer feasible. Despite increasing availability of some of these molecular features in most cancer centers, POLE mutation testing has not routinely been available, and as yet there are no algorithms to direct management based upon molecular status thus practice variability is large. A prospective trial will get all components of the molecular classifier into the hands of clinicians and patients. Investigators have evidence-based publications supporting treatment recommendations herein, although taken from retrospective series or preclinical work. Investigators have a randomized controlled trial in molecular classification-driven care (PORTEC4a) that although not mature enough to be published has revealed no concerns for higher rates of adverse events in the observation-only arms that would threaten continuation. As clinicians are already beginning to factor molecular features into their management recommendations it is imperative that investigators measure the impact of implementation of molecular based triage in a controlled setting. This will enable us to have preassigned 'stop' mechanisms in place if higher than anticipated recurrence rates are note and has the potential to change future algorithms for care.

NB: This trial will be conducted in compliance with the protocol, GCP and all applicable regulatory requirements.

Statistical design:

Primary Endpoint:

The primary aim of this study is to provide reliable estimates of the 3-year cumulative incidence of pelvic recurrence, and to confirm that this probability is sufficiently low e.g. de-escalation or no adjuvant therapy is safe in molecular classification selected early stage ECs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma, with one of the following combinations of FIGO stage, grade, and LVI: Stage IA (not confined to polyp), grade 3 (with or without LVI), pN0 Stage IB, grade 1, 2 pNx/N0 with or without LVI Stage IB, grade 3 without LVI pN0 Stage II (microscopic), grade 1 or 2, pN0 and without substantial LVI Surgery consisting of hysterectomy (total abdominal, laparoscopic or robotic-assisted) and bilateral salpingo-oophorectomy. Lymph node dissection can be performed as per institutional standards (sentinel or full lymphadenectomy). Pelvic LN assessment is required for grade 3 or stage II cancers. Para-aortic lymphadenectomy is not mandated.
* Age ≥18 years
* Eastern Cooperative Group (ECOG) performance status 0, 1 or 2.
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy for endometrial cancer or previous pelvic radiation.
* History of another invasive malignancy, except for non-melanoma skin cancers or tumors curatively treated with no evidence of disease for ≥ 5 years
* Inability to be registered and receive treatment within 12 weeks of hysterectomy .
* Abnormal p53 (p53abn) and/or mismatch repair deficiency (MMRd) on immunohistochemistry without pathogenic POLE mutation.
* MELF (microcystic, elongated and fragmented (MELF)) pattern of invasion is excluded within p53wt/NSMP tumors, not POLEmut

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Pelvic recurrence | every 6 months for the first 3 years
  recurrent disease in the pelvis (including the vagina)

SECONDARY OUTCOMES:
Recurrence free survival | every 6 months for the first 3 years
  duration of time from registration to time of relapse or death, whichever occurs first
Overall survival | every 6 months for the first 3 years
  duration of time from registration to time of death from any cause.
Sites of relapse | every 6 months for the first 3 years
  local (vagina), regional (pelvic and/or paraaortic nodal), or distant.
Patient Decisional Conflict Scale | through study completion, an average of 3 years
  a validated tool reflecting patient decision making prior to and post intervention or new information
Variation in treatment | through study completion, an average of 3 years
  proportion of cases enrolled where adjuvant treatment administered deviated from recommendations

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Vancouver Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided